CLINICAL TRIAL: NCT06695130
Title: A Phase 1/2, Parallel, Randomized, Modified Double-blind, Multi-arm Study to Assess the Safety and Immunogenicity of a Combination Vaccine Comprised of Different Recombinant Spike Antigen Levels of a Matrix-M Adjuvanted Recombinant COVID-19 Vaccine and Recombinant Influenza Vaccine in Adult Participants 50 Years of Age and Older
Brief Title: Study of a Combination Vaccine Comprised of Different Recombinant Spike Antigen Levels of a Matrix-M Adjuvanted Recombinant COVID-19 Vaccine and Recombinant Influenza Vaccine in Adult Participants 50 Years of Age and Older
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VBT00002
Record Dates: First submitted 2024-11-14; First posted 2024-11-19 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: COVID-19 Immunization; Influenza Immunization
Keywords: COVID-19 Vaccine; Influenza Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is modified double-blind:
  * Investigator, participants, and laboratory personnel will be blinded
  * Clinical site staff preparing/administering the study vaccines will be unblinded
  * Sponsor study staff will be blinded, except for dedicated staff involved in interim analysis, who will be unblinded at the time of interim analysis, and for dedicated staff involved in assessing criteria for safety surveillance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Group 1: RIV (in right or left deltoid) and placebo (in opposite deltoid) (Experimental): two IM injections on D01
  Interventions: Biological: RIV (recombinant influenza vaccine); Other: Placebo (0.9% NaCl)
- Group 2: rC19 (dose 1) (in right or left deltoid) and placebo (in opposite deltoid) (Experimental): two IM injections on D01
  Interventions: Biological: rC19 (dose 1); Other: Placebo (0.9% NaCl)
- Group 3: RIV (in right or left deltoid) and rC19 (dose 1) (in opposite deltoid) (Experimental): two IM injections on D01
  Interventions: Biological: RIV (recombinant influenza vaccine); Biological: rC19 (dose 1)
- Group 4: RIV + rC19 (dose 1) (in right or left deltoid) and placebo (in opposite deltoid) (Experimental): two IM injections on D01
  Interventions: Biological: RIV + rC19 (dose 1); Other: Placebo (0.9% NaCl)
- Group 5: RIV + rC19 (dose 2) (in right or left deltoid) and placebo (Experimental): two IM injections on D01
  Interventions: Biological: RIV + rC19 (dose 2); Other: Placebo (0.9% NaCl)
- Group 6: RIV + rC19 (dose 3) (in right or left deltoid) and placebo (Experimental): two IM injections on D01
  Interventions: Biological: RIV + rC19 (dose 3); Other: Placebo (0.9% NaCl)
- Group 7: RIV + rC19 (dose 4) (in right or left deltoid) and placebo (in opposite deltoid) (Experimental): two IM injections on D01
  Interventions: Biological: RIV + rC19 (dose 4); Other: Placebo (0.9% NaCl)

INTERVENTIONS:
Biological: RIV (recombinant influenza vaccine) — Influenza, inactivated, split virus or surface antigen
  Other Names: Recombinant influenza vaccine
  Arms: Group 1: RIV (in right or left deltoid) and placebo (in opposite deltoid); Group 3: RIV (in right or left deltoid) and rC19 (dose 1) (in opposite deltoid)
Biological: rC19 (dose 1) — Protein subunit
  Other Names: Novavax's adjuvanted recombinant COVID-19
  Arms: Group 2: rC19 (dose 1) (in right or left deltoid) and placebo (in opposite deltoid); Group 3: RIV (in right or left deltoid) and rC19 (dose 1) (in opposite deltoid)
Biological: RIV + rC19 (dose 1) — RIV component: Influenza, inactivated, split virus or surface antigen NVXC19 component: Protein subunit
  Arms: Group 4: RIV + rC19 (dose 1) (in right or left deltoid) and placebo (in opposite deltoid)
Biological: RIV + rC19 (dose 2) — RIV component: Influenza, inactivated, split virus or surface antigen NVXC19 component: Protein subunit
  Arms: Group 5: RIV + rC19 (dose 2) (in right or left deltoid) and placebo
Biological: RIV + rC19 (dose 3) — RIV component: Influenza, inactivated, split virus or surface antigen NVXC19 component: Protein subunit
  Arms: Group 6: RIV + rC19 (dose 3) (in right or left deltoid) and placebo
Biological: RIV + rC19 (dose 4) — RIV component: Influenza, inactivated, split virus or surface antigen NVXC19 component: Protein subunit
  Arms: Group 7: RIV + rC19 (dose 4) (in right or left deltoid) and placebo (in opposite deltoid)
Other: Placebo (0.9% NaCl) — Normal saline
  Arms: Group 1: RIV (in right or left deltoid) and placebo (in opposite deltoid); Group 2: rC19 (dose 1) (in right or left deltoid) and placebo (in opposite deltoid); Group 4: RIV + rC19 (dose 1) (in right or left deltoid) and placebo (in opposite deltoid); Group 5: RIV + rC19 (dose 2) (in right or left deltoid) and placebo; Group 6: RIV + rC19 (dose 3) (in right or left deltoid) and placebo; Group 7: RIV + rC19 (dose 4) (in right or left deltoid) and placebo (in opposite deltoid)

SUMMARY:
Study VBT00002 is planned to be a Phase 1/2, randomized, modified double-blind, active-controlled, multi-center study to be conducted in approximately 980 adults aged 50 years and older in the United States. The purpose of the study is to assess the safety and immunogenicity of recombinant influenza vaccine (RIV) + adjuvanted recombinant COVID-19 vaccine (rC19) vaccine comprised of RIV combined with different recombinant Spike (rS) antigen levels of rC19 compared to RIV alone, rC19 (dose 1) alone, and RIV and rC19 (dose 1) (coadministered in opposite arms). Placebo will be coadministered in the RIV alone, rC19 (dose 1) alone, and RIV + rC19 study groups to control for the number of injections and to maintain observer blinding. Thus, each participant will receive two injections at enrollment, one in each deltoid muscle.

Study details include:

* The study duration will be approximately 12 months
* Study intervention will be administered via a single intramuscular (IM) injection into the right and left deltoid muscles on Day(D) 01
* Dose escalation with sequential enrollment (sentinel cohort followed by main cohort for a given dose)
* The visit frequency for participants will be D01 and D30, and D09-D366 (telephone call)

Number of Participants:

Approximately 980 participants are expected to be randomized.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria to be checked at Screening Visit:

* Aged 50 years or older on the day of inclusion Informed consent
* Informed consent form has been signed and dated.
* Able to attend all scheduled visits and to comply with all study procedures.
* Participant must be able to receive an injection in the deltoid muscle of both arms.
* Participant must have completed a primary vaccination series against SARS-CoV-2 and at least 1 booster with a locally authorized or approved COVID-19 vaccine.

Inclusion criteria to be checked at Visit 1 (Day [D]01):

* Aged 50 years or older on the day of inclusions
* Participants who are healthy or with pre-existing stable condition (defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 12 weeks before enrollment), as determined by medical evaluation including medical history and physical examination.
* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

  * Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, or surgically sterile.

OR

• Is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to study intervention administration until at least 4 weeks after study intervention administration.

A female participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) on the day of enrollment before the first dose of study intervention.

* Informed consent form has been signed and dated.
* Able to attend all scheduled visits and to comply with all study procedures.
* Participant must be able to receive an injection in the deltoid muscle of both arms.
* Participant must have completed a primary vaccination series against SARS-CoV-2 and at least 1 booster with a locally authorized or approved COVID-19 vaccine.

Exclusion Criteria to be checked at Screening Visit and at Visit 1 (D01):

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (for glucocorticoids, ≥ 10 milligrams/day of prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known systemic hypersensitivity to any of the study intervention components, or history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances .
* Self-reported thrombocytopenia, contraindicating intramuscular injection, based on investigator's judgment.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular injection, based on investigator's judgment.
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion .
* Any illness that, in the opinion of the investigator, would pose a health risk to the participant if enrolled.
* Moderate or severe acute illness/infection (according to investigator judgment) or febrile illness (temperature ≥ 100.4°F) on the day of study intervention administration. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Alcohol, prescription drug, or substance abuse that, in the opinion of the Investigator, might interfere with the study conduct or completion.
* History of serious adverse reaction to any influenza or COVID-19 vaccines.
* Personal or family history of Guillain-Barré syndrome.
* Prior history of myocarditis, pericarditis, or myopericarditis.
* Prior history of stroke or stroke risk factors, which may include untreated/uncontrolled hypertension, hyperlipidemia, or diabetes; active smoking; obesity, based on investigator's judgment; history of thromboembolic disease; cardiac structural abnormality; atrial fibrillation; carotid stent placement; or family history of stroke.

Prior/concomitant therapy

* Receipt of any vaccine in the 4 weeks preceding study intervention administration or planned receipt of any vaccine prior to the second blood draw (ie, approximately in the 28 days following study intervention administration.
* Previous vaccination against influenza (in the previous 6 months) with an investigational or marketed vaccine.
* Previous vaccination against COVID-19 (in the previous 6 months) with an investigational or marketed vaccine OR history of COVID-19 in the previous 6 months.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 980 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-04-03 (Estimated); Study Completion 2026-04-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with immediate adverse events (AEs) | Immediate adverse events are any unsolicited systemic adverse events reported in the 30 minutes after vaccination
  Within the 30 minutes after vaccination
Number of participants with solicited injection site reactions | Up to 7 each days after vaccination
  Solicited injection site reactions include injection site pain, erythema and swelling
Number of participants with solicited systemic reactions | Up to 7 days after each vaccination
  Solicited systemic reactions include fever, headache, fatigue, myalgia and chills
Number of participants with unsolicited AEs | Up to 28 days after each vaccination
  Unsolicited (spontaneously reported) AEs, not fulfilling criteria for solicited adverse reactions
Number of participants with adverse events of special interest (AESIs) | Up to 180 days after each vaccination
  AESIs
Number of participants with medical attended adverse events (MAAEs) | Up to 180 days after each vaccination
  MAAEs
Number of participants with MAAEs relating to predefined PIMDs | From Day 182 through 12 months following the last study vaccination
  MAAEs relating to predefined PIMDs
Number of participants with serious adverse events (SAEs) | Up to 180 days after each vaccination
  SAEs
Number of participants with related SAEs | From Day 182 through 12 months following the last study intervention
  Related SAEs
Number of participants with MAAEs relating to predefined PIMDs that meet the criteria for SAEs | From Day 182 through 12 months following the last study vaccination
  MAAEs relating to predefined PIMDs that meet the criteria for SAEs
Geometric mean (GM) of HAI titers in all participants | At Day 01 and Day 30
  HAI titers
Geometric mean ratio (GMR) of HAI titers in all participants | At Day 01 and Day 30
  Individual HAI titers ratio Day 30/Day 01
GM of SARS-CoV-2 neutralizing titers in all participants | At Day 01 and Day 30
  SARS-CoV-2 neutralizing titers
GMR of SARS-CoV-2 neutralizing titers ratio D30/D01 in all participants | At Day 01 and Day 30
  Individual SARS-CoV-2 neutralizingtiters ratio Day 30/Day 01

SECONDARY OUTCOMES:
Percentage of participants with seroconversion in all participants | At Day 30
  Seroconversion is defined by:HAI titer < 10 [1/dil] at Day 01 and post-injection titer ≥ 40 [1/dil] at Day 30 or HAI titer ≥ 10 [1/dil] and a ≥ 4-foldincrease in titer [1/dil] at Day 30
Percentage of participants with HAI titer ≥ 10 (1/dil) in all participants | At Day 01 and Day 30
  detectable HAI titer ≥ 10 (1/dil)
Percentage of participants with HAI titer ≥ 40 (1/dil) in all participants | At Day 01 and Day 30
  HAI titer ≥ 40 (1/dil)
Percentage of participants with seroresponse to SARS-CoV-2 in all participants | At Day 30
  Seroresponse to SARS-CoV-2 isdefined by SARS-CoV-2 neutralizingtiters ≥ 4-fold rise in SARS-CoV-2neutralizing titers from Day 01 to Day 30

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Central Phoenix Medical Clinic- Site Number : 8400009, Phoenix, Arizona
  - Synexus Clinical Research US, Inc. - Cerritos- Site Number : 8400002, Cerritos, California
  - Synexus Clinical Research US - Vista- Site Number : 8400010, Vista, California
  - Optimal Research - Florida- Site Number : 8400006, Melbourne, Florida
  - Synexus Clinical Research US - Orlando- Site Number : 8400007, Orlando, Florida
  - Optimal Research - Illinois- Site Number : 8400008, Peoria, Illinois
  - Synexus Clinical Research US - Evansville- Site Number : 8400004, Evansville, Indiana
  - Walgreens Clinical Trials-Malden- Site Number : 8400012, Malden, Massachusetts
  - Synexus Clinical Research US - Minneapolis- Site Number : 8400011, Richfield, Minnesota
  - Synexus-Las Vegas- Site Number : 8400005, Las Vegas, Nevada
  - Synexus Clinical Research US - Cincinnati- Site Number : 8400003, Cincinnati, Ohio
  - Synexus Clinical Research US - Anderson- Site Number : 8400001, Anderson, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org